CLINICAL TRIAL: NCT06837246
Title: A Randomized, Parallel, Double-Blind, Placebo-Controlled Study to Assess Cognitive Effects of Cognitive Nutritional Supplementation in the General Population
Brief Title: A Clinical Trial to Assess Cognitive Effects of Cognitive Nutritional Supplement in General Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmavite LLC (Industry)
Collaborators: Balchem Corporation (Industry); Biofortis, Inc. (a Mérieux NutriSciences company) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-2409
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cognition; Concentration; Attention; Focus
Keywords: cognition; concentration; attention; problem-solving; capsule; clinical trial; placebo-controlled; focus; memory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Nutritional Supplement (Placebo Comparator): Intervention is pills of cognitive nutrient
  Interventions: Dietary Supplement: Cognitive Nutritional Supplement
- Placebo (Active Comparator): Intervention is pills of matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cognitive Nutritional Supplement — Pills of cognitive nutritional supplement
  Arms: Cognitive Nutritional Supplement
Other: Placebo — Matching placebo to active
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, 12-week parallel study that aims to determine the effects of a cognitive nutritional supplement for 12 weeks on cognition parameters specific to attention/focus related domains, compared to a placebo control, in a general population of adult men and women in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥25 to ≤65 years of age at screening.
2. English is the primary spoken language.
3. Able to operate a study-provided iPad connected to the internet with a strong and reliable internet connection.
4. Willing to consume 3 capsules per day for 12 weeks.
5. Willing to review and follow all training materials provided.
6. Willing to avoid alcohol, marijuana/hemp products (including CBD products), and vigorous physical activity 24 h prior to the baseline (week 0), mid-point (Week 6), and end of study (Week 12) cognition testing days.
7. Non-user or former user (cessation ≥12 months of screening) of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco, nicotine gums or lozenges) with no plans to begin use during the study period.
8. Willing to maintain habitual diet and physical activity patterns throughout the study.
9. Willing to refrain from exclusionary medications, supplements, and products throughout the study.
10. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Principal Investigator.

Exclusion Criteria:

Cognition related criteria

1. Diagnosed neurological disorder such as Alzheimer's disease, Parkinson's disease, stroke, intracranial hemorrhage, or any brain lesions including tumors.
2. Diagnosed mental health disorder, such as major depressive disorder or any anxiety disorder. The use of daily or as-needed prescription medications to treat these conditions is also exclusionary.
3. Any infective or inflammatory brain disease, including those of viral, fungal, or syphilitic etiologies.
4. Elective hospitalizations planned (e.g., elective cosmetic procedures) during the study period.
5. Color blindness or visual impairments that cannot be corrected with glasses or contact lenses.
6. Diagnosed sleep disorder (e.g., sleep apnea) or occupation where sleep during the overnight hours is irregular (e.g., 3rd shift of overnight workers).
7. History of repeated head injury (e.g., concussions from sports activities) or single trauma resulting in a period of unconsciousness lasting 1 h or more.
8. Diagnosis of a learning and/or behavioral disorders such as dyslexia.
9. Diagnosis of attention-deficit/hyperactivity disorder (ADHD).
10. Use of any dietary supplements, other than a conventional once-daily multivitamin/mineral supplement that does not contain certain nutrient with cognitive effects, during the study period. Participants will be allowed to discontinue use of exclusionary dietary supplements during the screening period.
11. Experienced a major life stress event, including the death of a loved one, marriage or divorce, birth of a child, unemployment, or moved to a new residence, within the last 6 months.

    General health related criteria
12. History or presence of cancer in the prior two years, except for non-melanoma skin cancer.
13. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and unwilling to commit to the use of a medically approved form of contraception throughout the study period.

    General safety related criteria
14. Exposure to any non-registered drug product or has participated in another intervention study within 30 days prior to screening.
15. Recent history (within 12 months of visit 1) of alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz. beer, 5 oz. wine, or 1½ oz. distilled spirits).
16. Another household member is a current participant in this study.
17. Any condition the Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

6.2.1 Excluded Products

* Tobacco / nicotine products within 12 months of screening and throughout the study period
* Any non-registered drug product within 30 days of screening
* Alcohol within 24 h of each cognition test day
* Marijuana/hemp products (including CBD products) within 24 h of each cognition test day
* Current use of any medication used to treat mental health disorders, such as major depressive disorder or any anxiety disorder
* Current use of any medications used to treat ADHD
* Current use of any dietary supplements, other than a conventional once-daily multivitamin/mineral supplement that does not contain certain nutrient with cognitive effect. Participants will be allowed to discontinue use of exclusionary dietary supplements during the screening period.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Feature Match | Week 0, Week 6, and Week 12
  Overall Score: The sum of the difficulties of all successfully answered problems, minus the sum of the difficulties of all incorrectly answered problems

SECONDARY OUTCOMES:
Feature Match | Week 0, Week 6, and Week 12
  Overall Reaction Time (ms): The average time taken to respond correctly
  Total Number of Errors: Sum of incorrect responses
SART Test | Week 0, Week 6, and Week 12
  Total Number of Errors: Sum of all commission errors (total count of inappropriate responses to a non-target stimulus [the number 3] and all omission errors (total number of times the participant failed to respond to a target stimulus [any number other than 3]
Double Trouble | Week 0, Week 6, and Week 12
  Overall Score: The number of correctly answered problems, minus incorrect ones
Spatial Span | Week 0, Week 6, and Week 12
  Overall Score (points): Total number of points scored during the task (points are awarded to each correctly solved puzzle, with more points awarded for more difficult puzzles)
Token Search | Week 0, Week 6, and Week 12
  Average Score (number of boxes): Average number of boxes in which all tokens were located without error
Rotations | Week 0, Week 6, and Week 12
  Overall Score: The sum of the difficulties of all successfully answered problems, minus the sum of the difficulties of all incorrectly answered problems
Number Ladder | Week 0, Week 6, and Week 12
  Maximum Level Completed: The hardest level (i.e., the problem with the highest number of targets) that the individual successfully completed
Paired Associates | Week 0, Week 6, and Week 12
  Maximum Level Completed: The hardest level (i.e., the problem with the highest number of targets) that the individual successfully completed
Odd One Out | Week 0, Week 6, and Week 12
  Overall Score: The number of correctly answered problems, minus incorrect ones
Polygons | Week 0, Week 6, and Week 12
  Overall Score: The sum of the difficulties of all successfully answered problems, minus the sum of the difficulties of all incorrectly answered problems
Grammatical Reasoning | Week 0, Week 6, and Week 12
  Overall Score: The number of correctly answered problems, minus incorrect ones
Digit Span | Week 0, Week 6, and Week 12
  Overall Score: The highest number completed
Spatial Spanning | Week 0, Week 6, and Week 12
  Overall Score: (The minimum number of moves required to solve the puzzle * 2) - (the number of moves actually made)
THAT | Week 0, Week 6, and Week 12
  Alertness rating (Sum of individual Likert scale scores)
Food Frequency Questionnaire: Total Kcal/Day | Week 0 and Week 12
  Healthy Eating Index (HEI)-2020: Total kcal/d
Food Frequency Questionnaire: Total carbohydrate (g/d) | Week 0 and Week 12
  Healthy Eating Index (HEI)-2020: Total carbohydrate (g/d)
Food Frequency Questionnaire: Total fiber (g/d) | Week 0 and Week 12
  Healthy Eating Index (HEI)-2020: Total fiber (g/d)
Food Frequency Questionnaire: Total fat (g/d) | Week 0 and Week 12
  Healthy Eating Index (HEI)-2020: Total fat (g/d)
Food Frequency Questionnaire: Total protein (g/d) | Week 0 and Week 12
  Healthy Eating Index (HEI)-2020: Total protein (g/d)
Food Frequency Questionnaire: Total intake of other essential nutrient (mg/d) | Week 0 and Week 12
  Healthy Eating Index (HEI)-2020: Total intake of other certain essential nutrient (mg/day)
Food Frequency Questionnaire: Total caffeine (mg/day) | Week 0 and Week 12
  Healthy Eating Index (HEI)-2020: Total caffeine (mg/day)

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No